CLINICAL TRIAL: NCT02240017
Title: Randomized, Multicenter, Phase II/III Study, Evaluating Fractionated Cisplatin Chemotherapy/Gemcitabine Versus Carboplatin/Gemcitabine in the Treatment of Advanced or Metastatic Urothelial Cancer With Impaired Renal Function.
Brief Title: A Study Evaluating Chemotherapy With Fractionated Cisplatin/Gemcitabine Versus Carboplatin/Gemcitabine in the Treatment of Advanced or Metastatic Urothelial Cancer With Impaired Renal Function.
Acronym: VEFORA
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Institut Claudius Regaud (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13 URO 02
Record Dates: First submitted 2014-09-05; First posted 2014-09-15 (Estimated); Last update posted 2019-08-09 (Actual); Status verified 2019-08

CONDITIONS: Advanced Urothelial Cancer; Metastatic Urothelial Cancer
Keywords: Urothelial cancer, renal function impaired.
MeSH Terms: interventions — Carboplatin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Carboplatin/Gemcitabine (Active Comparator)
  Interventions: Drug: Carboplatin; Drug: Gemcitabine
- Fractionated Cisplatin/Gemcitabine (Experimental)
  Interventions: Drug: Fractionated Cisplatin; Drug: Gemcitabine

INTERVENTIONS:
Drug: Carboplatin — Carboplatin AUC (area under curve) 4,5 at day 1 of each cycle until 6 cycles.
  Arms: Carboplatin/Gemcitabine
Drug: Fractionated Cisplatin — Cisplatin 35mg/m² at day 1 and day 8 of each cycle until 6 cycles.
  Arms: Fractionated Cisplatin/Gemcitabine
Drug: Gemcitabine — Gemcitabine 1000mg/m² at day 1 and day 8 of each cycle until 6 cycles.

SUMMARY:
This is a phase II/III, multicenter, randomized study which includes 420 patients on six years + 3 years follow up. 92 patients will be included during the phase II ; additional 328 patients will be included.

Patients with an advanced or metastatic urothelial cancer with impaired renal function will be randomized in one of the two following chemotherapy arm:

* Fractionated Cisplatin + Gemcitabine.
* Carboplatin + Gemcitabine.

The main objective of the part II study will be to evaluate the efficacy and the safety of a chemotherapy with a doublet platinum salt compound/Gemcitabine with fractionated Cisplatin or Carboplatin in this population.

The main objective of the part III study will be to compare the efficacy in terms of overall survival of a chemotherapy with a doublet platinum salt/Gemcitabine with fractionated Cisplatin or Carboplatin in this population.

ELIGIBILITY:
Inclusion Criteria:

1. . Age < or = 18 years, patients aged 75 years or more will benefit from a geriatric assessment.
2. . Advanced or metastatic urothelial cancer confirmed histologically or cytologically.
3. . Patients liable to receive a first -line chemotherapy for advanced or metastatic urothelial carcinoma.
4. . Measurable disease according to RECIST criteria V1.1.
5. . Patients who received neoadjuvant or adjuvant chemotherapy based on platinum salt must have completed treatment at least 6 months before entering the study.
6. . Performance status < or = 2.
7. . Life expectancy > 3 months.
8. . Patients with creatinine clearance between 40 and 60 ml / min ( according to Cockcroft and Gault ).
9. . Patients having no contra-indication to overhydration.
10. . Satisfactory hematological tests: Neutrophils > 1.5 G / l Platelets > 150 G / l , hemoglobin ≥ 10 g / dl.
11. . Satisfactory liver function tests: total bilirubin < 1.5 x ULN (upper limit of normal), AST (aspartate aminotransferase) and ALT (alanine aminotransferase)<or = 2.5 x ULN (or 5 x ULN if liver metastases).
12. . In case of prior radiotherapy, a minimum of 14 days must relapse between the end of radiotherapy and study entry.
13. . For women of childbearing age , use an effective contraceptive method to study entry and for the duration of the study and 6 months after the last dose of study treatment ; For sexually active fertile men having a partner of childbearing age using effective contraception for the duration of the study and 6 months after the last dose of study treatment.
14. . Patient affiliated to a social security system in France.
15. . Patient signed informed consent before inclusion in the study and before any specific procedure for the study.

Exclusion Criteria:

1. . Any concomitant or previous malignancy within 5 years prior to the study ( with the exception of basal cell or squamous cell carcinoma in situ).
2. . Pregnant or lactating women.
3. . Patients with brain metastases or meningeal or symptoms suggestive of such secondary locations.
4. . Bisphosphonate or Denosumab treatment initiated within 28 days prior to randomization into the study or patient who have started such treatment during the study ( a bisphosphonate or denosumab treatment initiated within a period longer than 28 days before randomization may be continued without change during the study ).
5. . Other concomitant cancer (radiation therapy, radiopharmaceutical agent chemotherapy).
6. . Patients with uncontrolled infection.
7. . Patients with peripheral neuropathy grade> 1, whatever the origin or patients with hearing loss.
8. . Patient with unstable disease (eg: unstable diabetes, poorly controlled hypertension , congestive heart failure or myocardial infarction within 3 months prior to study entry).
9. . Known hypersensitivity to study drugs.
10. . Treatment with any other investigational drug within 30 days before inclusion.
11. . Any psychological condition , familial, sociological or geographical not to comply with medical monitoring and / or procedures in the study protocol.
12. . Patient protected by law.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2015-01-21 (Actual); Primary Completion 2018-04-10 (Actual); Study Completion 2019-07-15 (Actual)

PRIMARY OUTCOMES:
Phase II: Efficacy - Rate of non progression at the end of treatment (C6D21). | 5 years.
  Progression is defined according to RECIST (Response Evaluation Criteria in Solid Tumors) criteria V1.1.
Phase III: Overall survival (in months). | 9 years.
  Overall survival is defined as the time from randomization until death or last follow up news (censured data).
Phase II: Tolerance - Percentage of patients for whom at least one of the 3 defined tolerance criteria (see description) is observed. | 5 years.
  Defined tolerance criteria :
  * Postponement of chemotherapy > or = 2 weeks.
  * Alteration of renal function.
  * Need to decrease twice Gemcitabine dose on day 1 for : NCI CTC (National Cancer Institut Common Toxicity Criteria) grade III or IV non-hematologic toxicity, hematologic toxicity.

SECONDARY OUTCOMES:
Phase II and III: Objective response. | Phase II: 5 years ; Phase III: 9 years.
  Objective response (ie complete or partial response) will be evaluated according to RECIST v1.1 criteria.
Phase II and III: Tolerance according to NCI toxicity scale (version 4.0). | Phase II: 5 years ; Phase III: 9 years.
Phase II and III: Geriatric evaluation using questionnaires. | Phase II: 5 years ; Phase III: 9 years.
  The geriatric assessment will be evaluate using the following questionnaires: G8 (oncodage) , ADL (activity of daily living), CIRSG (cumulating illness rating scale geriatric) , MMS (mini-mental score), IADL (instrumental activities of daily living), GDS (geriatric depression scale), MNA (mini-nutritional assessment).
Phase II and III: Quality of life using the EORTC QLQ - C30 questionnaire (European Organization for research and treatment of Cancer - Quality of life questionnaire). | Phase II: 5 years ; Phase III: 9 years.
Phase II and III: Pharmacokinetics - Platin concentrations | At cycles 1 and 2 day 1 - 5 mn before the end of infusion, one hour after the end of infusion, 3 hours (arm A) or 4 hours (arm B) after the end of infusion.
Phase II and III: Pharmacogenetics, exploration of cytidine deaminase activity and study of its genetic polymorphisms. | Prior to the initial dose on cycle 1 day 1.
Phase II and III: Progression free survival. | Phase II: 5 years ; phase III: 9 years.
  Progression free survival will be evaluated according to RECIST v1.1 criteria.
Phase II and III: Overall survival. | Phase II: 5 years ; Phase III: 9 years.
  Overall survival is defined as the time from randomization until death from all causes combined.
Phase II and III: Time to treatment failure. | Phase II: 5 years ; Phase III: 9 years.
  Time to treatment failure is defined as the time from randomization to treatment discontinuation, whatever its cause.

CONTACTS AND LOCATIONS:
Overall Officials: Loic MOUREY, MD, Study Chair — Institut Claudius Regaud
Locations (18):
- France (18):
  - INSTITUT DE CANCEROLOGIE DE L'OUEST - Site Paul Papin, Angers
  - Chru Besancon - Hopital Jean Minjoz, Besançon
  - Institut Bergonie, Bordeaux
  - Centre Francois Baclesse, Caen
  - Centre Georges Francois Leclerc, Dijon
  - CH VERSAILLES - Hôpital André Mignot, Le Chesnay
  - CHU LIMOGES - Hôpital Dupuytren, Limoges
  - Centre Leon Berard, Lyon
  - Institut Paoli Calmettes, Marseille
  - Ch Mont de Marsan, Mont-de-Marsan
  - Institut Regional Du Cancer Montpellier, Montpellier
  - Ap-Hp-Hopital Saint-Louis, Paris
  - INSTITUT DE CANCEROLOGIE DE L'OUEST - Site René Gauducheau, Saint-Herblain
  - Institut de Cancerologie Lucien Neuwirth, Saint-Priest-en-Jarez
  - CHU de STRASBOURG, Strasbourg
  - Institut Claudius Regaud, Toulouse
  - Chru Tours, Tours
  - Institut Gustave Roussy, Villejuif